CLINICAL TRIAL: NCT06381752
Title: Value of Continuous Passive Motion in Rehabilitation After Total Knee Replacement - A Prospective Randomized Controlled Multicenter Trial.
Brief Title: Value of Continuous Passive Motion in Rehabilitation After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Erol Gercek, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CPMvsPT
Record Dates: First submitted 2024-04-05; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Total Knee Arthroplasty
Keywords: CPM; inpatient rehabilitation; Staffelstein Score
MeSH Terms: interventions — Motion Therapy, Continuous Passive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in inpatient rehabilitation randomly assigned to this group Assigned intervention: CPM the (Other): Invervention group
  Interventions: Device: Continuous passive motion
- Patients in inpatient rehabilitation randomly assigned to this group Assigned intervention: group p (Other): Control group
  Interventions: Other: standard rehabilitation

INTERVENTIONS:
Device: Continuous passive motion — Daily application of continuous passive motion
  Arms: Patients in inpatient rehabilitation randomly assigned to this group Assigned intervention: CPM the
Other: standard rehabilitation — standard rehabilitation program with group physiotherapy
  Arms: Patients in inpatient rehabilitation randomly assigned to this group Assigned intervention: group p

SUMMARY:
Immediate rehabilitation after total knee arthroplasty (TKA) differs in terms of volume, intensity but also type of treatment. Continuous passive motion after TKA is so far only investigated for replacing physiotherapy. This study is conducted to investigate CPM when it partially replaces group physiotherapy in terms of functional and patient-reported outcomes.

DETAILED DESCRIPTION:
The aim of this study is to analyze the value (knee function, pain, and quality of life) of continuous passive motion (CPM) after total knee replacement (TKR), when it partially replaces group physiotherapy (PT) in inpatient rehabilitation to save human resources. Patients are randomized to CPM group, consisting of 3 daily sessions of 20 minutes each, or to group PT, consisting of 25 minutes physiotherapy in groups 5 days weekly. Multimodal rehabilitation does not differ for both groups throughout the 3-week rehabilitation stay.

Primary outcome is the Staffelstein Score, German standard score in rehabilitation. Secondary outcomes are Oxford Knee Score (OKS), active and passive range of motion (ROM), and pain on visual analogue scale (VAS). Return to work is assessed by post-operative days.

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty because of knee osteoarthritis
* Inpatient rehabilitation in participating clinics

Exclusion Criteria:

* Pregnancy
* Not able to give informed consent
* Psychological disorders
* Body weight > 150 kg
* Hip range of motion < 50°

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Staffelstein Score | baseline (t0) and 3 weeks later (t1)
  A maximum score of 120 points is possible including 3 sub dimensions with a maximum score of 40 points each. Sub dimensions consist of pain, activities of daily life (ADL), and ROM. The Staffelstein Score is assessed by a professional investigator. Higher scores indicated better results.

SECONDARY OUTCOMES:
Oxford Knee Score (OKS) | baseline (t0), 10 days after baseline (t1), 3 weeks after baseline (t2), 4 months after baseline (t3)
  Assessing patient's functional status. A maximum score of 48 points is possible including 12 questions with 0 - 4 points for each question [12]. Higher scores indicated better functional outcomes.
Range of motion (ROM) | baseline (t0), 10 days after baseline (t1), 3 weeks after baseline
  Range of motion (ROM): Assessing the patient's knee range of motion with a mechanical goniometer
Visual Analogue Scale (VAS) | baseline (t0), 10 days after baseline (t1), 3 weeks after baseline (t2)
  The patient rates pain during rest and during movement and draws a vertical line on a 10cm line with 0 cm indicating no pain and 10 cm indicating maximum pain
Return to work | baseline (t0), 4 months after baseline (t3)
  Assessed by post-operative days until first day of work

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaetsmedizin der JGU Mainz, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No